CLINICAL TRIAL: NCT04694911
Title: Development of the Oncology Opportunity Cost Assessment Tool (OOCAT)
Brief Title: Development of the Oncology Opportunity Cost Assessment Tool
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 19G.854; JT 14788 (Other: JeffTrial Number)
Record Dates: First submitted 2020-12-07; First posted 2021-01-05 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Focus Groups; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health Services Research (focus group, interview, OOCAT): FOCUS GROUP: Patients participate in focus group session over 60-90 minutes.
  COGNITIVE INTERVIEW: Patients complete cognitive interview on the clarity, interpretability, and ease of use of the OOCAT.
  FEASIBILITY TESTING: Patients receive OOCAT at the point of care, online, or via telephone, per patients' preference.
  Interventions: Behavioral: Focus Group; Other: Interview; Other: Research or Clinical Assessment Tool

INTERVENTIONS:
Behavioral: Focus Group — Participate in focus group
Other: Interview — Complete cognitive interview
Other: Research or Clinical Assessment Tool — Receive OOCAT
  Other Names: Clinical Assessment Tool, Clinical Assessment Tool, Clinical or Research Assessment Tool

SUMMARY:
This study develops and tests an instrument to measure opportunity costs called the Oncology Opportunity Cost Assessment Tool (OOCAT) in cancer patients. Patients experience significant costs, both direct financial as well as indirect costs, associated with seeking cancer treatment. While the direct financial impact of care on patients is receiving increased attention, other important consequences, such as opportunity cost, remain largely unmeasured. Opportunity cost is an economics term that refers to the loss of potential benefits from other options when one option is chosen - if resources are used for one purpose, they are no longer available for the next best option. The information and knowledge gained from this study may help researchers develop the OOCAT, which may allow them to understand the opportunity cost of treatment for each patient. The OOCAT may then be used to determine not just the best medications for patients, but also the best comprehensive treatment plan that will allow them to get the right treatment in the right place at the right time.

ELIGIBILITY:
Inclusion Criteria:

* Treated for cancer at one of the 3 participating sites (Jefferson Center City, Jefferson Methodist Hospital, Jefferson Abington)
* English speaking
* Able to attend and participate in a focus group

Exclusion Criteria:

* Treated at a Jefferson site other than the ones mentioned
* Non-English Speaking

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Patients treated for cancer at Jefferson Center City, Jefferson Methodist Hospital, or Jefferson Abington
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Patient-level opportunity costs associated with oncology care | 1 Day of Interview
  Patient-identified themes that contribute to opportunity cost will be generated via patient focus groups
Development of the Oncology Opportunity Cost Assessment Tool (OOCAT) | 1 Day of Interview
  Will organize themes into domains and will generate items representing each of the themes for inclusion in an instrument designed to measure patient opportunity cost of seeking care. Will perform cognitive interviews with a random sampling of patients from the cancer center to test initial instrument items to ensure content validity and clarity of each item.
Implementation of OOCAT | 1 Day of OOCAT administration
  Will test the instrument as developed with patients receiving oncology care across the Jefferson Health System to gather preliminary data informing the reliability of the scale to measure opportunity cost of seeking care.

CONTACTS AND LOCATIONS:
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States